CLINICAL TRIAL: NCT03407261
Title: OHRQoL Assessment Between Sliding Anterior Retraction and Micro-osteoperforations for Accelerated Orthodontics in Patients Who Were Assigned for Pre-molar Extraction and Decompensation
Brief Title: OHRQoL and Accelerated Orthodontics With Micro-osteoperforations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, LIANA FATTORI ABATI, PhD student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Fattori3
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micro-osteoperforations (Experimental): Minimally invasive micro-osteoperforations procedure used to achieve accelerated orthodontic tooth movement. Topical and local anesthetic will be delivered in the area to be treated in accordance with standard practice
  Interventions: Procedure: micro-osteoperforations
- Control (No Intervention): Anterior retraction after premolars extraction will be done conventionally (sliding mechanics)

INTERVENTIONS:
Procedure: micro-osteoperforations — Three vertical micro-osteoperforations, using Excellerator, in the buccal extracted site were executed following the aseptic procedure and local anesthesia
  Arms: Micro-osteoperforations

SUMMARY:
OHRQoL assessment using OHIP-14 between sliding anterior retraction with self-ligating brackets and micro-osteoperforations for accelerated orthodontics in orthognathic surgery patients who were assigned for pre-molar extraction and decompensation

DETAILED DESCRIPTION:
Our patients are participants in a randomized clinical trial, an ongoing study about the effectiveness of micro-osteoperforations to accelerate tooth movement. The study sample consisted of 22 consecutive subjects - 12 females and 10 males - between the ages of 18 and 35, who were selected for ortho-surgical treatment and pre-molar extraction assigned for decompensation. The participants were randomly allocated to two groups: control (anterior retraction was performed using implant-assisted sliding mechanics with self-ligating brackets) and experimental (micro-osteoperforations were performed in the activation appointments for anterior retraction using implant-assisted sliding mechanics). For immediate and follow-up assessment of patients' perceptions, comparing regular orthodontic activation and activation with Accelerated Orthodontics, subjects were asked to complete an electronic questionnaire OHIP-14, to assess the participants' comfort level, experiences, and QoL impact.

ELIGIBILITY:
Inclusion Criteria:

* maxillomandibular discrepancy indicative for orthognathic surgery, no previous dental extractions, good oral and general health, non-smokers, and no use of systemic corticosteroids or biphosphonates

Exclusion Criteria:

* any tooth absence/previous tooth extraction

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-10-21 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Comparision of OHRQoL between groups - OHIP-14A | 4 days
  comparision of OHIP-14A results between groups after appointment for anterior retraction: The sum of the numeric scores for each participant in all 14 items, with a maximum score of 56 (4x14);
Comparision of OHRQoL between groups - 7 domains | 4 days
  comparision of each OHIP-14 domain results between groups after appointment for anterior retraction: To evaluate which domains had the most impact during the trial, the answers for each question were combined as pairs and summed for statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- FOUSP, São Paulo, Brazil